CLINICAL TRIAL: NCT05282875
Title: Evolution of Anti-HLA Immunization According to Immunosuppressive Therapy Management Modalities in Kidney Transplant Patients Returning to Dialysis in Lorraine Between January 2007 and December 2019
Brief Title: Anti-HLA Immunization And Immunosuppressive Therapy Management In Kidney Transplant Patients Returning to Dialysis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GIRERD Sophie, MD, PhD, Central Hospital, Nancy, France
Other Study IDs: 2021PI192
Record Dates: First submitted 2022-03-08; First posted 2022-03-16 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Kidney Transplantation; Immunosuppressive Agents; HLA Sensitization; Dialysis
Keywords: immunosuppressive agents; graft loss; HLA antibodies; retransplantation; kidney transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- kidney transplant patients returning to dialysis after graft loss: This cohort contains kidney transplant patients returning to dialysis after graft loss in Lorraine between 1 January 2007 and 31 December 2019. They are identified by the REIN registry of the Lorraine region.
  The REIN registry is a national database that contains multiple information on patients with chronic end-stage renal disease (type of nephropathy, type of replacement therapy, comorbidities).
  Interventions: Drug: management of immunosuppressive therapy

INTERVENTIONS:
Drug: management of immunosuppressive therapy — 3 groups :
  * Discontinuation of immunosuppressive agents
  * Reduction of immunosuppressive agents
  * Maintenance of immunosuppressive agents

SUMMARY:
This study is an analytical observational retrospective cohort study. It is a single-center study conducted in the Nancy University Hospital.

End stage renal disease is the ultimate stage of the chronic kidney disease. Patients need extra-renal replacement techniques. Kidney transplantation is the most effective option for survival, quality of life and costs.

Then long-term immunosuppressive agents are required to prevent allograft rejection and improve graft survival.

The number of patients who return in dialysis after graft loss is increasing and accounts for 10% of incident dialysis patients and 14% of patients on the kidney transplant waiting list registered in 2019. This population may develop complications induced by end-stage renal disease and adverse events related to prolonged exposure to immunosuppressive agents.

There are currently no formal guidelines on the management of immunosuppressive agents when patients return to dialysis. Reduction or discontinuation of therapy appears to decrease cardiovascular, infectious, and neoplastic complications. However, continuing these treatments may limit anti-HLA sensitization which may access to retransplantation.

Only a few low-powered cohort studies have evaluated the impact of the management of immunosuppressive therapy on the HLA-sensitization.

The hypothesis of our study is that the continuation of immunosuppressive agents when patients return in dialysis may limit anti-HLA sensitization. Therefore, access to retransplantation could be facilitated.

The main objective is to compare the evolution of anti-HLA sensitization according to the management of immunosuppressive treatment after the return in dialysis (maintenance, reduction, cessation).

Secondary objectives are time to re-transplantation for patients on the transplant waiting list, survival of the new graft, patient survival, and dialysis complications (cardiovascular, infectious and neoplastic complications).

DETAILED DESCRIPTION:
Cohort constitution :

The cohort of patients returning to dialysis after graft loss is extracted from the REIN (Réseau Epidémiologique et Information en Néphrologie) Lorraine registry, which follow all patients in end-stage renal failure under replacement therapy in the Lorraine region since 2001.

Patients returning to dialysis after graft loss between 1st January 2007 and 31st December 2019 are extracted from the register and included.

From this cohort, 3 groups were created according to the management of their immunosuppressive therapy : maintenance, reduction, and discontinuation. The immunological data of the patients are recovered from the HLA laboratory of the Nancy University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the Lorraine regional REIN registry over the period 2007-2019,
* Returning in dialysis after a kidney transplantation, with a living or deceased donor.
* On haemodialysis or peritoneal dialysis.
* Registered or not on the waiting-list for retransplantation

Exclusion Criteria:

* Patients with graft dysfunction receiving a pre-emptive retransplantation
* Absence of serum tested for anti-HLA (human leukocyte antigen) antibodies after the return to dialysis.
* No information on immunosuppressive agents

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The cohort of patients returning to dialysis after graft loss is extracted from the REIN Lorraine registry. Patients returning in dialysis after graft loss between 1st January 2007 and 31st December 2019 are included.
  From this cohort, 3 groups were created according to the management of their immunosuppressive therapy : maintenance, reduction, and discontinuation. The immunological data of the patients are recovered from the HLA laboratory of the Nancy University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the evolution of anti-human leucocyte antigen sensitization according to the management of immunosuppressive therapy | baseline = return in dialysis, t1=6 months after return in dialysis
  Evolution of the panel reactive antibody evolution 6 months after the return in dialysis

SECONDARY OUTCOMES:
Patients survival | baseline = return in dialysis, end of follow up = death or last follow-up or 31 december 2020
  Patient survival after return in dialysis
New transplantation | baseline = return in dialysis, end of follow up = death or last follow-up or 31 december 2020
  Retransplantation after return in dialysis
Graft Survival after retransplantation | baseline = return in dialysis, end of follow up = death or last follow-up or 31 december 2020
  Graft Survival after retransplantation
Incidence of infectious, neoplastic and cardiovascular events | baseline = return in dialysis, end of follow up = 1 year after return in dialysis
  Incidence of infection, neoplastic and cardiovascular events after return in dialysis

CONTACTS AND LOCATIONS:
Locations (1):
- Central HNF, Nancy, Lorraine, France

IPD SHARING:
Plan to Share IPD: No